CLINICAL TRIAL: NCT03865381
Title: Onduo Virtual Diabetes Clinic Study
Acronym: VDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 100901
Record Dates: First submitted 2019-02-25; First posted 2019-03-06 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Virtual Diabetes Clinic (Other): The Onduo Virtual Diabetes Clinic (VDC) is the suite of diabetes management services including remote monitoring, diet/lifestyle coaching, medication management accessed via Onduo App and partner apps. Subjects will engage with a Care Lead through the App and will have a medical consultation via telemedicine with an Onduo VDC Physician.
  Interventions: Device: Onduo App

INTERVENTIONS:
Device: Onduo App — The Onduo App is a software application which tracks data relevant to diabetes care, such as, but not limited to, medication, meal logs and glucose readings, and activity data. The Onduo App connects wirelessly to a Care Team Console through the Internet. The Onduo App may also connect wirelessly to commercially available FDA-regulated (i.e., cleared and approved) medical devices and non-medical devices through the subject's Smartphone.

SUMMARY:
This is a prospective, single arm study designed to evaluate the change in hemoglobin A1c after 4 months of participation in the Onduo Virtual Diabetes Clinic (VDC) in individuals with Type 2 diabetes and suboptimal glycemic control.

DETAILED DESCRIPTION:
The Onduo Virtual Diabetes Clinic (VDC) is the suite of diabetes management services accessed via a software application (Onduo App).

Eligible subjects are asked to use the Onduo App and commercially available FDA-regulated medical devices and non-medical devices, for up to 4 months.

Subjects receive a continuous glucose monitor (CGM) and are asked to use the device for up to 6 wear cycles of 10 days each.

Subjects are scheduled for a medical review via a face-to-face telemedicine consultation with a VDC Physician.

Subjects may have their diabetes medications changed by a VDC Physician following their telemedicine visit.

Information provided to a subject in the course of the study is not intended as a substitute for the subject's primary care provider's guidance.

At the completion of the subject's study participation, the Onduo App will be deactivated and there will be no further data collection through the app.

A1c levels and surveys are collected at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female; 18 years of age or older
* Confirmed diagnosis of Type 2 diabetes mellitus
* Willing to use CGM and BGM
* A1c result ≥8.0% and ≤12.0%
* Receive their diabetes care from Premier Medical Associates or the Palo Alto Medical Foundation
* Own a Smartphone with a data plan and be the primary user of that smartphone
* Smartphone must use a supported Android OS or iOS

Exclusion Criteria:

* Pregnant or breastfeeding
* Use of an insulin pump
* Any condition or situation that the Sponsor or Investigator determines as inappropriate for study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Majithia, MD, Principal Investigator — Onduo
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation, Palo Alto, California
  - Premier Medical Associates, Monroeville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Majithia AR, Erani DM, Kusiak CM, Layne JE, Lee AA, Colangelo FR, Romanelli RJ, Robertson S, Brown SM, Dixon RF, Zisser H. Medication Optimization Among People With Type 2 Diabetes Participating in a Continuous Glucose Monitoring-Driven Virtual Care Program: Prospective Study. JMIR Form Res. 2022 Apr 5;6(4):e31629. doi: 10.2196/31629. PMID 35147501
- [Derived] Majithia AR, Kusiak CM, Armento Lee A, Colangelo FR, Romanelli RJ, Robertson S, Miller DP, Erani DM, Layne JE, Dixon RF, Zisser H. Glycemic Outcomes in Adults With Type 2 Diabetes Participating in a Continuous Glucose Monitor-Driven Virtual Diabetes Clinic: Prospective Trial. J Med Internet Res. 2020 Aug 28;22(8):e21778. doi: 10.2196/21778. PMID 32856597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Diabetes Clinic
Started | 60
Completed | 55
Not Completed | 5
Not completed — Protocol Violation/Non-Compliance | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35
  Asian | 9
  Black or African American | 6
  Other | 4
  White, American Indian or Alaska Native, Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  No, not of Hispanic, Latino/a, or Spanish origin | 51
  Yes, of Hispanic, Latino/a, or Spanish origin | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55
Weight [Mean (Standard Deviation); unit: lb] | 218.7 (59.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.7 (7.2)
HbA1c [Mean (Standard Deviation); unit: Percent (%)] | 8.9 (1.0)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 132.1 (15.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.7 (10.4)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 168.3 (42.8)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 40.4 (9.1)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 100.1 (36.5)
Non-HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 128.0 (42.70)
Total Cholesterol/HDL Ratio [Mean (Standard Deviation); unit: Ratio] | 4.4 (1.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 236.7 (194.3)
Diabetes Medications [Count of Participants; unit: Participants]
  0 | 0
  1 | 6
  2 | 21
  >=3 | 28
Type of Diabetes Medications [Count of Participants; unit: Participants]
  Alpha glucosidase inhibitor | 1
  Biguanide | 46
  DPP-4 inhibitor | 10
  GLP-1 analogue | 14
  Insulin | 20
  SGLT2 inhibitor | 20
  Sulfonylurea | 30
  Thiazolidinedione | 2
  Lipid-lowering medications | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin A1c
Description: Mean change in hemoglobin A1c from enrollment to 4 months
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 55
Percent (%) | -1.6 (1)

2. Secondary Outcome: Change in Weight From Enrollment
Description: Change in weight from enrollment to 4 months
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 54
lb | -9.0 (10.4)

3. Secondary Outcome: Time to First Change in Diabetes Medication or Dosage From Enrollment
Description: Change in diabetes medication or dosage from enrollment
Time Frame: 4 Months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Mean Glucose From the First Wear Period Versus the Final Wear Period.
Description: Mean glucose was calculated from an initial wear period to a final wear period.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 43
mg/dL | -14.6 (27.5)

5. Secondary Outcome: Change in Glycemic Variability From the First Wear Period Versus the Final Wear Period.
Description: Coefficient of variation was calculated from an initial wear period to a final wear period.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 43
Percent (%) | -1.6 (4.5)

6. Secondary Outcome: Change in Time Spent in Glycemic Range From the First Wear Period Versus the Final Wear Period.
Description: Percent time in Glycemic Range, 70 to 180 mg/dL, was calculated from an initial wear period to a final wear period.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Virtual Diabetes Clinic
Number analyzed (Participants) | 43
Percent (%) | 10.2 (20.5)

7. Secondary Outcome: Mean Change in A1c
Description: Mean change in estimated A1c between the first and second CGM wear periods, where estimated A1c is a linear function of average blood glucose.
Time Frame: 4 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Virtual Diabetes Clinic
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03865381/Prot_SAP_000.pdf